CLINICAL TRIAL: NCT07047027
Title: Microbial Communities in Root Canal Infections of Patients With Diabetes.
Brief Title: Comparative Analysis of Root Canal Microbiota in Diabetic and Systemically Healthy Patients
Status: Completed | Type: Observational
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Sevinç Aktemur Türker, Professor, Bulent Ecevit University
Other Study IDs: 2024-27194235-03
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Root Canal Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — root canal contents
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study was to assess the influence of Diabetes Mellitus on the microbial flora involved in root canal infections through a comparative analysis with that of systemically healthy patients.

DETAILED DESCRIPTION:
A total of 39 participants aged 18 to 65 years were enrolled in the study, including 21 patients with Diabetes Mellitus and 18 systemically healthy individuals (controls). In the diabetic group, 12 teeth were diagnosed with persistent endodontic infections (SEI) and 9 with primary endodontic infections (PEI). In the healthy group, 12 teeth presented with SEI and 6 with PEI. Root canal samples were obtained using sterile paper points, transferred into Eppendorf tubes containing phosphate-buffered saline (PBS), and stored at -80 °C until analysis. The V3-V4 hypervariable regions of 16S rRNA from both sample types were amplified and sequenced using the Illumina MiSeq platform. Amplicon sequence variants (ASVs), generated via the DADA2 pipeline, were analyzed in the QIIME2 environment and taxonomically assigned using the SILVA database. Microbial richness and diversity were assessed using alpha diversity indices (Chao1, Shannon, Simpson, Faith's PD, Fisher alpha) and beta diversity metrics (Bray-Curtis, Jaccard, Unweighted UniFrac, and Weighted UniFrac). Alpha and beta diversity metrics were compared using the Kruskal-Wallis test and pairwise permutational multivariate analysis of variance (PERMANOVA), respectively, via the phyloseq package in R (version 4.1). Differentially abundant taxa were identified using Linear Discriminant Analysis Effect Size (LEfSe).

ELIGIBILITY:
Inclusion Criteria:The inclusion criteria for patient selection were as follows: patients in the diabetic group were required to have a diagnosis of type 2 Diabetes Mellitus with no other systemic diseases; patients in the control group had to be systemically healthy with no history of any systemic illness. All participants must not have used antibiotics within the past three months, must not be pregnant, and must have teeth with intact coronal restorations that prevent direct pulp exposure to the oral environment. Only asymptomatic teeth diagnosed with chronic apical periodontitis and a Periapical Index (PAI) score of 3 or higher were included -

Exclusion Criteria:The exclusion criteria were: teeth with extensive coronal destruction that would prevent rubber dam isolation, presence of pain, swelling, or sinus tract, presence of root or crown fractures, and periodontal pockets deeper than 3 mm.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who were attended to the faculty of dentistry
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-02-21 (Actual); Study Completion 2025-03-13 (Actual)

PRIMARY OUTCOMES:
Microbial analysis | 8 weeks
  Root canal microbial flora

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry of Bulent Ecevit University, Zonguldak,, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No